CLINICAL TRIAL: NCT00486174
Title: Intermittent Bolus Infusion of Methylene Blue to Reduce Norepinephrine Requirements in Sepsis: A Randomized Controlled Trial
Brief Title: Methylene Blue in Sepsis: A Randomized Controlled Trial
Acronym: SMURF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: primary site withdrew due to competing study: never enrolled any subjects.
Sponsor: Queen's University (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Dr. Daniel W Howes, Queen's University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMED-090-07; PSI Grant application #2006-36
Record Dates: First submitted 2007-06-12; First posted 2007-06-14 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2008-05

CONDITIONS: Sepsis
Keywords: Sepsis; Methylene Blue; Norepinephrine
MeSH Terms: conditions — Sepsis | interventions — Methylene Blue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): standard sepsis therapy plus Methylene Blue
  Interventions: Drug: methylene blue
- 2 (No Intervention): standard sepsis therapy

INTERVENTIONS:
Drug: methylene blue — 2.0 mg/kg of Methylene Blue administered every 6 hours (as required) for up to 48 hours.
  Arms: 1

SUMMARY:
The purpose of this study is to investigate whether the addition of Methylene Blue to the standard treatment of septic shock will reduce vasopressor requirements

DETAILED DESCRIPTION:
The management of severe infections, sepsis and septic shock is a serious problem facing physicians. Septic shock kills 10,000 Canadians every year. It is the most common cause of death in intensive units and the rates of sepsis and septic shock continue to increase annually.

Septic shock is a complex interaction between pathologic vasodilation, relative and absolute hypovolemia, myocardial depression, and altered microvascular function resulting from a systemic inflammatory response to infection. After restoration of the circulating volume, many patients continue to suffer from a maldistribution of blood flow. Current hypotheses suggest that global indicators of hypoperfusion (serum lactate, hypotension, decreased oxygen delivery) represent an averaging of areas of normal or increased blood flow with areas where blood flow is decreased. These under-perfused areas become more hypoxic. The resulting tissue damage leads to more inflammation and more maldistribution, perpetuating a vicious cycle progressing on to death.

Vasopressive agents are used in an attempt to maintain mean arterial blood pressure and restore perfusion, but these agents work globally, potentially worsening blood flow to the under-perfused areas. As well, many vasopressors have deleterious side effects such as metabolic and endocrine functions, and changes to regional blood flow.

The microvascular changes are mediated by primarily nitric oxide (NO). Baseline levels of nitric oxide are produced by constitutive Nitric Oxide Synthase (cNOS), with NO levels measured in the nano-molar range. Inflammatory mediators cause increased production of inducible Nitric Oxide Synthase (iNOS) leading to NO levels measured in the micro-molar range.

Suppression of nitric oxide production using non-specific NOS inhibitors has had discouraging results. Methylene Blue is a selective iNOS inhibitor. The purpose of this pilot study is to confirm safety and demonstrate signs of benefit in the use of methylene blue in sepsis. In particular, this study will examine whether the addition of methylene blue to standard early goal directed therapy in sepsis will reduce vasopressor requirements.

ELIGIBILITY:
Inclusion Criteria:

* First presentation of sepsis syndrome: clinical evidence of infection with Systemic Inflammatory Response Syndrome (SIRS)as defined by two or more of:

  * Temperature > 38°C or < 36°C,
  * Heart rate > 90 beats per minute,
  * One or more of respiratory rate > 20, hyperventilation with PaCO2 < 32 mm Hg, requiring mechanical ventilation,
  * One or more of white blood cells > 12,000 X 109 /L or white blood cells < 4000 X 109 /L or immature neutrophils > 10%.
* Undergoing early goal directed therapy with a mean arterial blood pressure (MAP) < 65 mmHg despite fluid resuscitation to CVP > 10mmHg.
* Able to provide informed consent as per our institutional standard.
* To receive first dose of study drug within six hours of first recorded hypotension (MAP < 65mmHg).

Exclusion Criteria:

* Age < 18 years.
* Undergoing palliation.
* Not expected to survive 48 hours.
* Resuscitated from a vital sign absent arrest.
* Ongoing dialysis.
* Anuric or creatinine > 300 μmol/L.
* Pregnant.
* Patient or family history of glucose-6-phosphate dehydrogenase deficiency.
* Allergic to methylene blue, phenothiazines, thiazide diuretics, or food dyes.
* Patient mass > 150 kg.
* Demonstrated Pulmonary Hypertension (Mean Pulmonary Artery Pressure > 25 mmHg by Swan Ganz Catheter or Echo demonstrated Right Ventricular Systolic Pressure > 40 mmHg).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-06

PRIMARY OUTCOMES:
The primary outcome of interest is to assess the norepinephrine requirements in the methylene blue groups to maintain a mean arterial blood pressure greater or equal to 65 mmHg in comparison to the control group. | hourly for 96 hours

SECONDARY OUTCOMES:
safety of methylene blue | 96 hours
survival to ICU discharge | 30 days
survival to hospital discharge | 30 days
total norepinephrine administered | 96 hours
number of whole hours norepinephrine free | hourly for 96 hours

CONTACTS AND LOCATIONS:
Overall Officials: Daniel W Howes, MD, Principal Investigator — Queen's University